CLINICAL TRIAL: NCT06933199
Title: Neoadjuvant Stereotactic Radiotherapy for Brain Metastasis - Prospective Trial NeoSTROBE
Brief Title: Neoadjuvant Stereotactic Radiotherapy for Brain Metastasis
Acronym: NeoSTROBE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: University Hospital Olomouc (Other); Masaryk Memorial Cancer Institute (Other); University Hospital Hradec Kralove (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONK-NeoSTROBE; NW25-03-00278 (Other Grant/Funding Number: Ministry of Health of the Czech Republic)
Record Dates: First submitted 2025-04-03; First posted 2025-04-18 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Brain Metastases
Keywords: Brain Metastases; Neoadjuvant Stereotactic Radiotherapy; Leptomeningeal Disease; Quality of Life; Overall Survival; Acute Toxicity
MeSH Terms: conditions — Brain Neoplasms; Meningeal Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will include two groups of study subjects, enrolled prospectively and analysed retrospectively
Masking Description: No masking will be used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant NaSRT - prospective (Experimental): Patients undergoing neoadjuvant NaSRT will be enrolled prospectively in this study arm.
  Interventions: Radiation: Neoadjuvant Stereotactic Radiotherapy (NaSRT)
- Postoperative SRT - retrospective (Active Comparator): Patients who underwent postoperative SRT in the past will be analyzed retrospectively in this study arm.
  Interventions: Radiation: Postoperative Stereotactic Radiotherapy (SRT)

INTERVENTIONS:
Radiation: Neoadjuvant Stereotactic Radiotherapy (NaSRT) — Neoadjuvant Stereotactic Radiotherapy (NaSRT) gives radiotherapy before surgery from many different angles around the body. The beams meet at the tumor. This means the tumor receives a high dose of radiation and the tissues around it receive a much lower dose. This lowers the risk of side effects.
  Arms: Neoadjuvant NaSRT - prospective
Radiation: Postoperative Stereotactic Radiotherapy (SRT) — Postoperative Stereotactic Radiotherapy (SRT) gives radiotherapy after surgery from many different angles around the body. The beams meet at the tumor. This means the tumor receives a high dose of radiation and the tissues around it receive a much lower dose. This lowers the risk of side effects.
  Arms: Postoperative SRT - retrospective

SUMMARY:
This multicentre proof-of-concept study, involving 4 centers, aims to establish the value of fractionated neoadjuvant stereotactic radiotherapy (NaSRT) as a new treatment paradigm for brain metastases (BM) in the frame of the Czech neurooncology network. Most relevant studies published to date used single-fraction radiotherapy and dealt with the inherent bias related to their retrospective nature. The researchers aim to increase the level of evidence for this treatment paradigm together with other similar ongoing studies.

DETAILED DESCRIPTION:
The prospective study will evaluate the efficacy and toxicity of neoadjuvant stereotactic radiotherapy (NaSRT) in patients with brain metastases (BM). Clinical data gathered will include local control (LC), the incidence of leptomeningeal disease (LMD), radiological and clinical signs of radiation necrosis (RN), overall survival, and incidence of metachronous brain metastases. The magnetic resonance imaging (MRI) characteristics of irradiated and subsequently resected BM will be obtained according to the usual protocol and specified time intervals. Clinical monitoring will comprise neurological findings, Karnofsky performance status, and quality of life (FACT-Br/EORTC QLQ-C30 questionnaire and EORTC QLQ-BN20 questionnaire. These questionnaires are designed to measure cancer patients' physical, psychological, and social functions. The questionnaires are composed of multi-item scales and single items). The data obtained from the retrospective control group (estimated for 160 patients) will include the same parameters monitored in the consecutive group of patients who underwent surgery at centers included in our study, with or without adjuvant radiotherapy (RT). Formation of this control group corresponding to the NaSRT group will enable the efficacy and risks of NaSRT to be determined in comparison with established treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Karnofsky Performance Status ≥ 60
* Histologically verified primary cancer disease
* MRI findings indicating BM
* Target BM indicated for surgical resection and any other metastases suitable for radical SRT.
* Target BM between 1 cm and 7 cm at the longest diameter on T1 post-contrast MR imaging

Exclusion Criteria:

* Confirmed hematological malignity
* Small-cell (lung) carcinoma
* Peracute condition requiring immediate neurosurgical intervention
* History of whole-brain radiotherapy (WBRT)
* History of stereotactic radiotherapy to a target brain metastasis
* Pregnancy
* Inability to perform surgical resection of the target BM within 7 days after NaSRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute Toxicity | 3 months
  Acute Toxicity will be assessed in the study subjects according to Common Terminology Criteria for Adverse Events (CTCAE) ver. 5 to 10%.
Quality of Life Questionnaire (FACT-Br/EORTC QLQ-C30) | 3 months
  Quality of Life will be assessed in the study subjects using the FACT-Br/EORTC QLQ-C30 questionnaire.
Quality of Life Questionnaire (EORTC QLQ-BN20) | 3 months
  Quality of Life will be assessed in the study subjects using the EORTC QLQ-BN20 questionnaire.

SECONDARY OUTCOMES:
Time from NaSRT to local progression | 3 years
  Time from NaSRT to local progression will be assessed.
Time from NaSRT to detection of LMD | 3 years
  Time from NaSRT to detection of LMD will be assessed.
Time from NaSRT to the onset of RN | 3 years
  Time from NaSRT to the onset of RN will be assessed.
Time from NaSRT to detection of distant parenchymal metastasis | 3 years
  Time from NaSRT to detection of distant parenchymal metastasis will be assessed.
Overall Survival | 3 years
  Overall survival from NaSRT to death from any reason will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Cvek, Assoc.Prof., MD, Ing, PhD, MBA, Principal Investigator — University Hospital Ostrava
Locations (4):
- Czechia (4):
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - Masaryk Memorial Cancer Institute, Brno
  - University Hospital Hradec Králové, Hradec Králové
  - University Hospital Olomouc, Olomouc

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] DeAngelis LM, Delattre JY, Posner JB. Radiation-induced dementia in patients cured of brain metastases. Neurology. 1989 Jun;39(6):789-96. doi: 10.1212/wnl.39.6.789. PMID 2725874
- [Background] CHAO JH, PHILLIPS R, NICKSON JJ. Roentgen-ray therapy of cerebral metastases. Cancer. 1954 Jul;7(4):682-9. doi: 10.1002/1097-0142(195407)7:43.0.co;2-s. No abstract available. PMID 13172684
- [Background] Gavrilovic IT, Posner JB. Brain metastases: epidemiology and pathophysiology. J Neurooncol. 2005 Oct;75(1):5-14. doi: 10.1007/s11060-004-8093-6. PMID 16215811
- [Background] Barnholtz-Sloan JS, Sloan AE, Davis FG, Vigneau FD, Lai P, Sawaya RE. Incidence proportions of brain metastases in patients diagnosed (1973 to 2001) in the Metropolitan Detroit Cancer Surveillance System. J Clin Oncol. 2004 Jul 15;22(14):2865-72. doi: 10.1200/JCO.2004.12.149. PMID 15254054
- [Background] Linskey ME, Andrews DW, Asher AL, Burri SH, Kondziolka D, Robinson PD, Ammirati M, Cobbs CS, Gaspar LE, Loeffler JS, McDermott M, Mehta MP, Mikkelsen T, Olson JJ, Paleologos NA, Patchell RA, Ryken TC, Kalkanis SN. The role of stereotactic radiosurgery in the management of patients with newly diagnosed brain metastases: a systematic review and evidence-based clinical practice guideline. J Neurooncol. 2010 Jan;96(1):45-68. doi: 10.1007/s11060-009-0073-4. Epub 2009 Dec 4. PMID 19960227